CLINICAL TRIAL: NCT04347044
Title: The Effect of Pulmonary Rehabilitation on Bronchoscopic Volume Reduction Process Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principle investigator, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLVR_PR
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-04

CONDITIONS: Emphysema; Pulmonary Rehabilitation; Bronchoscopic Lung Volume Reduction
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation Group (Experimental): Optimal medication and clinical follow-up plus Pulmonary rehabiltation
  Interventions: Other: Pulmonary Rehabilitation; Other: Standart care
- Non-Pulmonary Rehabilitation Group (Active Comparator): Optimal medication and clinical follow-up
  Interventions: Other: Standart care

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Exercise training+ Optimal medication and clinical follow-up
  Arms: Pulmonary Rehabilitation Group
Other: Standart care — Optimal medication and clinical follow-up

SUMMARY:
The data of patients undergoing bronchoscopic volume reduction procedure will be analyzed retrospectively. Patients will be divided into two groups as patients with and without Pulmonary Rehabilitation before the procedure, and changes in functional levels of patients will be compared.

DETAILED DESCRIPTION:
The data of patients who underwent bronchoscopic volume reduction between January 2013 and March 2019 will be examined.

Patients will be divided into two groups as pulmonary rehabilitation applied (PR group) and not applied (Control group) before the procedure.

Changes in the parameters of initial and rehabilitation follow-up will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75
* Patients with a diagnosis of emphysema and bronchoscopic procedures

Exclusion Criteria:

• Patients who develop complications related to the procedure after bronchoscopic procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Six minute walking test | 20 minutes
  The test was conducted in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Patients were asked to walk as far as they can. Prior to and following the test, oxygen saturation, heart rate and Borg fatigue rating were measured, and the walking distance were recorded
Pulmonary Function Tests | 15 minutes
  PFTs were performed by using the Sensormedics model 2400 (Yorba Linda, CA, USA) spirometry device, and according to the American Thoracic Society (ATS) guidelines

SECONDARY OUTCOMES:
Carbonmonoxide diffusion test | 15 minutes
  It will performed in the pulmonary function test laboratory using Cosmed Quark PFT (USA) with single-breath technique

IPD SHARING:
Plan to Share IPD: Undecided